CLINICAL TRIAL: NCT03119337
Title: Reducing Provider Workload While Preserving Patient Safety: A 2-Way Texting Intervention in Zimbabwe's Voluntary Medical Male Circumcision Program
Brief Title: Text-based Follow-up in Zimbabwe's Voluntary Medical Male Circumcision Program
Acronym: 2WT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Medic Mobile (Industry); International Training and Education Center for Health (Unknown); ZICHIRe (Unknown); University of Zimbabwe (Other)
Responsible Party: Principal Investigator, Caryl Feldacker, Clinical Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001839
Record Dates: First submitted 2017-03-31; First posted 2017-04-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Voluntary Medical Male Circumcision
Keywords: male circumcision, text-based follow-up, Zimbabwe,

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a prospective, un-blinded, randomized control trial (RCT) among VMMC clients in a 1:1 ratio of control to intervention. Study participants and clinic staff are not masked to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-based VMMC follow-up (Experimental): Follow-up conducted via daily text not through mandatory in person visits. Men may elect to come to the clinic if concerned about any complications but have no routine, scheduled follow-up visits.
  Interventions: Other: Text-based follow-up
- Routine VMMC follow-up care (No Intervention): Routine VMMC follow up care with in person visits according to national guidelines.

INTERVENTIONS:
Other: Text-based follow-up — 2wT clients will receive automated daily texts from days 1-14. If a 2wT VMMC client responds that he suspects an AE, a VMMC nurse will exchange modifiable, scripted texts with clients to determine symptoms, frequency, and severity. Then, if deemed necessary, the client will be asked to return to clinic the following day or earlier. If 2wT patients do not respond to texts on Day 2 or Day 7, the same MoHCC tracing process will be activated, after which they will be considered LTFU. All study participants will be asked to come to the clinic for study-specific, Day 14 follow-up to review healing and verify adverse event reporting. At Day 42, we will implement a brief text-based survey with 2wT clients to ascertain complete healing, providing stronger inferences at study completion.
  Arms: Text-based VMMC follow-up

SUMMARY:
Voluntary medical male circumcision (VMMC) in sub-Saharan Africa is safe: the average rate of moderate and severe adverse events (AEs) at the country level is 0.8%, corresponding to 99% of men healing without incident. To reach the global target of 20 million by 2018, VMMC productivity needs to double in countries already plagued by severe healthcare worker shortages like Zimbabwe. The ZAZIC consortium partners with the Zimbabwe Ministry of Health and Child Care (MoHCC) and performed over 120,000 VMMCs. Current VMMC care in Zimbabwe requires in-person, follow-up visits at post-operative days 2,7, and 42. Over 95% adhere to multiple follow-up visits within 14 days of VMMC. ZAZIC's program has an overall AE rate of 0.4%; therefore, overstretched clinic staff conducted more than 200,000 unnecessary reviews for VMMC clients without complications. High mobile phone ownership, severe healthcare worker shortages, and rapid VMMC scale up make ZAZIC's VMMC program an ideal setting to test a mobile health (mHealth) intervention to reduce provider workload while safeguarding patient safety. Through an un-blinded, prospective, randomized, control trial (RCT) in high-volume facilities providing VMMC, ZAZIC will implement an interactive, two-way texting (2wT) intervention to identify men healing without complication, allowing them to decline routine in-person follow up visits. 2wT will simultaneously identify men with any sign of an adverse event, encouraging rapid in-person follow-up when an AE is suspected on any day, reducing unnecessary visits while maintaining quality care. We aim to 1) determine if 2wT can safely reduce VMMC follow-up visits; 2) estimate the cost savings associated with 2wT over routine VMMC follow-up; and 3) assess the acceptability and feasibility of 2wT for further scale-up. It is expected that this intervention with be as safe as routine care while providing distinct advantages in terms of efficiency, costs, and reduced healthcare worker burden. This approach is innovative as it focuses on using a low-cost mHealth intervention to reduce provider workload without deterioration in quality care. The success of this intervention could lead to adoption of this intervention at the national level, increasing efficiency of VMMC scale up and reducing burdens on providers and patients

DETAILED DESCRIPTION:
The investigators propose to maintain patient safety while reducing the substantial VMMC follow-up workload burden by using two-way mobile phone texts to provide in-person review only for men who indicate a desire or need for follow-up. This tailored approach to post-procedure VMMC care could reduce unnecessary visits and remove barriers for VMMC clients without deterioration of quality care. ZAZIC's diverse, expert team of researchers from the University of Washington, Seattle, USA; the University of Zimbabwe; Medic Mobile, Nairobi, Kenya; and Zimbabwean partner organizations will test this mHealth intervention. The investigators believe that bi-directional, interactive, text-based short message service (SMS) during the most critical 14 days after circumcision will help men identify and act on any sign of an adverse event, thereby seeking in-person follow-up only when an AE is suspected and reducing unnecessary visits. Reduced in-person follow-up could also free healthcare workers to perform additional VMMC surgeries. Using a prospective, randomized control trial (RCT), our intervention compares two groups of clients with cell phones: 1) standard care (control group) and 2) clients who receive and respond to a daily text with in-person follow-up only if desired or if an AE is suspected (intervention). Both arms complete a study-specific, Day 14, in-person, follow-up review for verification of self-reports (intervention) and comparison (control). Our specific aims are to:

Aim 1: Determine if 2-way texting can safely reduce VMMC follow-up visits Approach: Un-blinded, prospective, non-inferiority, RCT in high-volume facilities providing VMMC. Two-way texting (2wT) will provide interactive, text-based follow-up. 2wT men healing without complication could decline in-person follow-up; those with suspected AEs will be referred to in-person care. The investigators will compare the safety outcome of combined moderate or severe AE rate ≤ Day 14 post-VMMC and the workload outcome of average number of in-person follow-up visits between control and intervention arms.

Aim 2: Estimate the cost savings associated with 2wT over routine VMMC follow-up Approach: The investigators will determine the programmatic costs of 2wT from a systems perspective, including the technology [24], healthcare worker costs, and client perspective. The investigators will estimate the incremental intervention costs relative to standard practice to quantify gains in healthcare efficiency for scale-up and adoption.

Aim 3: Assess the acceptability and feasibility of 2wT for further scale-up Approach: Qualitative interviews with VMMC healthcare workers and brief quantitative interviews with 2wT clients inform intervention acceptance. Meetings with local researchers and collaborators will further assess feasibility, adaptation, open-source collaborative development, and system integration for replication and sustainability in Zimbabwe and the region.

APPROACH Study overview: Following usability testing with both healthcare workers and 2wT VMMC clients, The investigators will test if two-way texting (2wT) reduces unnecessary follow-up visits without compromising patient safety (Aim 1) using a randomized control trial in large, urban VMMC clinics. The investigators will assess the costs of 2wT from technology, healthcare worker, and client perspectives to determine the costs incurred by MoHCC if adopted for scale-up (Aim 2). The investigators will assess acceptability and feasibility working towards system integration and sustainability in Zimbabwe and beyond (Aim 3).

Aim 1: Technology overview: Studies that demonstrate the impacts of mHealth interventions too often have evaluated technologies that are made 'from scratch' and as a result are not robust enough to merit widespread replication [48, 74]. By partnering with a well-established non-profit mHealth organization, Medic Mobile (http://medicmobile.org/), and integrating with their existing software platform, open-source community and current efforts to integrate with existing health information systems (HIS) throughout sub-Saharan Africa, our team and proposed intervention are well positioned to scale up and sustain any promising results. Since 2008, Medic Mobile has been a leader in the global mHealth community [75-77], equipping more than 13,500 health workers serving over 8 million people across 23 countries. The Mobile Medic Toolkit is an Android-based application that supports texting in any language and works with or without internet connectivity on basic phones, smartphones, tablets, and computers [78]. The existing, well-proven, app-based Toolkit that will be the basis for 2wT provides an automated and prioritized list of upcoming tasks, guiding health worker through actions (e.g., response waiting, referral). The Toolkit provides real-time progress indicators such as texting delivery rates and response rates. Data from mobile users are replicated to Medic Mobile web app and analytics tools for real-time response. The platform is highly configurable, currently supporting evidence-backed workflows and program implementation related to ensuring safe deliveries [79], tracking tuberculosis patients [80], boosting immunization rates [81] and monitoring stocks of essential medicines [82]. These adaptable tools are free, open-source, and developed using human-centered design with input from people delivering care in the hardest-to-reach communities. While this technology has never been used in a VMMC program and requires adaptation of the clinical content, the existing 2wT software toolkit already contains the robust messaging features discussed in this proposal (Figure 2). The software adaptation process to alter and test alternative clinical content and the local specifications requires little additional software development. The adaptation process will be completed by co-investigator, Holeman, with additional technical and training support provided by Nairobi-based technical experts.

Study sites and population: In Zimbabwe, 81% of people already had mobile phone subscriptions in 2014 [83], indicating that the technology infrastructure exists and uptake is high. 2wT will be implemented in existing VMMC sites in the Chitungwiza District, a district purposefully selected for its high VMMC volume clinic locations. Chitungwiza District, a suburb of Harare, has an estimated 300,000 eligible, HIV-negative men ages 15-29; only 14% of eligible men have been circumcised to date. The investigators will implement 2wT in up to 5 ZAZIC VMMC sites in Chitungwiza, sites averaging 50-200 VMMC/month. About 80% of VMMC clients are surgical, rather than PrePex device-based, clients.

Study preparation: The investigators will conduct a rapid situation analysis with healthcare workers, VMMC clients, and stakeholders to assess suitable responses to VMMC client texts, setting standards for text responses and in-person follow-up. The investigators will modify existing usability surveys for this public health context. A small pilot with 50 VMMC clients will include usability testing with both 2wT clients and nurses implementing the 2wT system, illuminating system experiences from both perspectives. Usability results will inform in-box modification, message format preferences (SMS or WhatsApp) and optimal message delivery (timing, frequency, language preferences). Experience from study coordinator and other team members will add detail to inform 2wT adaptation and modification of Standard Operating Procedures before implementation. The investigators will examine local infrastructure (e.g. electricity and cell network), and explore 2wT cost reduction options (e.g., text bundling, free-call back numbers) and adapt accordingly

Standard VMMC care (Control arm): ZAZIC follows all MoHCC protocols based on WHO guidelines [20] including routine surgical VMMC follow-up on post-surgery days 2, 7 and 42 (Table 1). Patients may seek care outside scheduled visits for suspicion of AEs at any healthcare facility at any time but most often return to their VMMC site. Referral cards for VMMC clients provide local numbers for patients to text, call, or request a call back for emergencies. A standardized approach is used to assess, identify, and record the severity of AEs [51]. All VMMC care, from assessment of all AEs through complete healing, is provided free to clients from MoHCC. Clients who do not return to the clinic for follow-up on Day 2 or Day 7 are traced: 3 attempts by phone and then up to 3 attempts at in-person tracking after which they are considered lost to follow-up (LTFU) [52]. There is no tracing for Day 42 visits. For the purposes of this study, control arm VMMC clients will be asked to come in on Day 14 for an additional follow-up visit. No active follow-up is provided at Day 14.

VMMC care procedures (2wT arm): The investigators will conduct a prospective, un-blinded, randomized control trial (RCT) among VMMC clients in a 1:1 ratio of control to intervention. Study participants and clinic staff are not masked to treatment. Men in the 2wT will receive routine VMMC surgical care and counseling, including referral cards for emergencies. 2wT clients will receive automated daily texts from days 1-14 (Table 1 and Figure 3). It is free to receive call and texts; it costs $0.05 to send a SMS in Zimbabwe [84]. If they respond that they suspect no adverse event, no immediate follow-up action will be taken. If a 2wT VMMC client responds affirmatively to any daily text that he suspects an AE, a VMMC nurse will exchange modifiable, scripted texts with the client to determine the symptoms, frequency, and severity. Then, if deemed necessary, the client will be asked to return to clinic the following day or earlier if an emergency is suspected. AE management will adhere to MoHCC standard care. If 2wT patients do not respond to texts on Day 2 or Day 7, the same MoHCC tracing process will be activated, after which they will be considered LTFU. All study participants will be asked to come to the clinic for study-specific, Day 14 follow-up to review healing and verify adverse event reporting. Day 14 was chosen for verification because 95% of all AEs within the ZAZIC VMMC program are reported Day 14 or earlier [50], suggesting that most AEs have occurred by this time point. In a previous field study of AEs, the most common AEs of bleeding and infection were found a mean of 6.7 and 9.0 days, respectively, after VMMC [29], further supporting the 14 day period used in this and a previous study[5]. The Day 14 review will be conducted by routine VMMC providers according to MoHCC review guidelines. At Day 42, The investigators will implement a brief text-based survey with 2wT clients to ascertain complete healing, providing stronger inferences at study completion.

ELIGIBILITY:
Inclusion: For health care workers (Aim 3):

1. are employees posted at the site;
2. are at least 18 years of age or over;
3. provide health care services to patients as part of the VMMC programs; and
4. are able to provide written informed consent.

For VMMC clients (Aims 1): Eligibility criteria for VMMC clients are:

1. 18 years or older;
2. possession of own phone at enrollment;
3. provides contact details (phone, physical location);
4. receives surgical VMMC;
5. willing to follow MoHCC VMMC protocols;
6. willing to come in Day 14;
7. Able and willing to respond to a questionnaire administered by phone 42 days after circumcision.

Exclusion for Healthcare workers:

1. not willing to participate
2. not willing to be recorded

Exclusion for VMMC clients:

1. men without cell phones;
2. those who chose PrePex as PrePex requires a device-removal visit 7 days after placement and has distinctly different follow-up protocols;
3. men who have an inter-operative AE during routine VMMC will be withdrawn from the study as these men will have known, additional follow-up risks and mandatory in-person visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men will be enrolled in the study on male circumcision. Health care workers may be male or female
Enrollment: 780 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Cumulative adverse event (AE) rate (moderate or severe) | ≤ Day 14 for each participant with analysis completed in year 1.
  Incidence of AEs before Day 14 will be extracted from routine VMMC data for both 2wT and control. Incident AEs on Day 14 will be identified, classified, and graded for severity using routine MoHCC protocols [26] and recorded on routine VMMC AE forms. The investigators will compare cumulative rates of any moderate or severe AE ≤ Day 14 between groups using Fisher's exact test as the expected number of AEs is low. The rates will be calculated per arm as: (# moderate + severe AEs)/(total # VMMC clients who attend 2, 7 or 14 Day follow-up visit). Multivariate logistic regression models (any AE v none) will quantify the magnitude of difference, adjusting for any potential confounders.
Mean number of in-person visits | Before 42 day visit for each participant with analysis completed in year 1.
  To determine follow-up visit reduction, the investigators will compare the mean number of in-person visits for intervention and control using a t-test. A multivariate linear regression model will further quantify the effect of intervention on visit reduction, adjusting for potential confounders.
2wT costs | The costing data collection will be completed by April 2018 at the completion of all study participant follow-up. Analysis will conclude in year 1
  The investigators will calculate the relative costs and outcomes (effects) of intervention versus control, including costs for technology, healthcare worker time, and client considerations (travel, text costs, missed work). The investigators will conduct both activity-based costing from the implementation perspective and from the technology perspective to extrapolate results as costs that would be incurred by the MoHCC should they elect widespread scale up of 2wT.
2WT acceptability | The acceptability activities will be completed by April 2018 at the completion of all study participant follow-up with analysis to commence after that point. Analysis will conclude in year 1.
  2wT acceptability, using study recruitment and enrollment logs in addition to the texting database, the investigators will describe levels of acceptance, participation, refusal and drop-out. The investigators will carry out key informant interviews (KIIs) with up to 8 health care workers to gauge acceptability, satisfaction, identify facilitators and barriers to program success, and ascertain suggestions for intervention improvement. KIIs will be audio recorded and transcribed. The investigators will also implement questionnaires at the Day 14 visit with a subset of 100 2wT VMMC clients to gauge satisfaction, estimate direct and indirect costs (time away from work, transportation costs), and ascertain suggestions for intervention improvement.
2WT feasibility | The feasibility activities be completed by April 2018 at the completion of all study participant follow-up with analysis to commence after that point. Analysis will conclude in year 1.
  For feasibility, costing data will be combined with usability and acceptability information.

SECONDARY OUTCOMES:
AE rates on Day 14 | Day 14 data collection for each participant with analysis to be completed in year 1.
  AE rates on Day 14
severity of AEs. | Day 14 data collection for each participant with analysis to be completed in year 1.
  severity of AEs.
time between 2wT AE text reporting and follow-up | Day 14 data collection for each participant with analysis to be completed in year 1.
  time between 2wT AE text reporting and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Caryl Feldacker, PhD, MPH, Principal Investigator — University of Washington
Locations (5):
- Zimbabwe (5):
  - 1. Chitungwiza Central Hospital, Chitungwiza, Stand Number 12096 Batanai ROAD Zengeza 4
  - 2. South Medical Citimed Chitungwiza Hospital, Chitungwiza, Stand Number 14656 Zengeza 4
  - 5. Seke North Clinic, Seke North, Stand Number: 16106 UNIT G
  - 4. Seke South Clinic, Seke South, Stand Number: 19188 UNIT L
  - Zengeza 3 Clinic, Chitungwiza, Stand Number: 7723 Cheuka WAY Zengeza 3

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Feldacker C, Holeman I, Murenje V, Xaba S, Korir M, Wambua B, Makunike-Chikwinya B, Holec M, Barnhart S, Tshimanga M. Usability and acceptability of a two-way texting intervention for post-operative follow-up for voluntary medical male circumcision in Zimbabwe. PLoS One. 2020 Jun 16;15(6):e0233234. doi: 10.1371/journal.pone.0233234. eCollection 2020. PMID 32544161
- [Derived] Feldacker C, Murenje V, Holeman I, Xaba S, Makunike-Chikwinya B, Korir M, Gundidza PT, Holec M, Barnhart S, Tshimanga M. Reducing Provider Workload While Preserving Patient Safety: A Randomized Control Trial Using 2-Way Texting for Postoperative Follow-up in Zimbabwe's Voluntary Medical Male Circumcision Program. J Acquir Immune Defic Syndr. 2020 Jan 1;83(1):16-23. doi: 10.1097/QAI.0000000000002198. PMID 31809358
- [Derived] Feldacker C, Murenje V, Barnhart S, Xaba S, Makunike-Chikwinya B, Holeman I, Tshimanga M. Reducing provider workload while preserving patient safety via a two-way texting intervention in Zimbabwe's voluntary medical male circumcision program: study protocol for an un-blinded, prospective, non-inferiority, randomized controlled trial. Trials. 2019 Jul 23;20(1):451. doi: 10.1186/s13063-019-3470-9. PMID 31337414